CLINICAL TRIAL: NCT01352013
Title: The Impact of Omega-3 Fatty Acid Supplements on Fibromyalgia (FM) Symptoms: A Randomized, Double-blind, Placebo-controlled Exploratory Study.
Brief Title: The Impact of Omega-3 Fatty Acid Supplements on Fibromyalgia Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Yoram Shir (Other)
Collaborators: McGill University (Other)
Responsible Party: Sponsor-Investigator, Dr. Yoram Shir, Doctor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Omega3-MGH
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Omega-3; Chronic Pain; Fatigue; Mood; docosahexaenoic acid (DHA); eicosapentaenoic acid (EPA)
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Fatigue | interventions — Docosahexaenoic Acids; Oils; Fatty Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colored olive oil (Placebo Comparator)
  Interventions: Dietary Supplement: Fatty Acids (placebo)
- Omega-3 (oil) (Active Comparator)
  Interventions: Dietary Supplement: Omega-3 (oil)

INTERVENTIONS:
Dietary Supplement: Omega-3 (oil) — 5ml daily with breakfast for 56 days.
  Other Names: NutraSea HP
  Arms: Omega-3 (oil)
Dietary Supplement: Fatty Acids (placebo) — 5ml daily with breakfast for 56 days.
  Arms: Colored olive oil

SUMMARY:
The purpose of this study is to find out if omega-3 fatty acid supplements are more effective than an inactive placebo at reducing pain, reducing fatigue and elevating mood in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65.
* A diagnosis of FM according to the American College of Rheumatology classification criteria(Wolfe et al., 1990)
* Negative urine pregnancy test at enrolment and willingness not to become pregnant for the duration of the study.
* Pain levels of at least 4 on 10-cm VAS at the time of recruitment.
* Ability to communicate in English or in French.
* Willing to sign an informed consent.
* If the patient is taking medication or natural health product (excluding omega-3 containing products) to treat fibromyalgia, she must be on a stable regimen for a minimum of two weeks before recruitment and be willing to keep this stable medication or natural health product regimen throughout the study period.
* If the patient is using other therapies to treat fibromyalgia such as TENS, acupuncture, exercise, psychotherapy, massage, physiotherapy, etc, she must be doing so for a minimum of two weeks before recruitment and be willing to continue those therapies throughout the study period.

Exclusion Criteria:

* Use of anticoagulants (Coumadin® or Plavix®), having a bleeding disorder or being scheduled for a surgical procedure. This is because omega-3 fatty acids can prolong bleeding time, although doses we propose to use are safe (see Risks section)
* Allergy to fish, olive oil, medium chain triglycerides, lemon, green tea, vitamin E or tylenol
* Past (within the last year) or present specific dietary supplementation with omega-3 fish oil or other natural health products containing omega-3 fatty acids (e.g. flax seed oil, krill oil, etc) or regularly eating more than two fatty fish meals/week (salmon, mackerel, sardine, flounder, herring, or any other fish considered to have a high level of omega-3 fatty acids).
* Patient enrolled in another research study involving any treatment.
* Patient engaged in active litigation
* Regular use of recreational drugs
* Alcohol consumption > 10 units/week
* Morbidly obese patients
* Pregnancy or breastfeeding
* Uncontrolled major medical conditions. Neurological problems. Current psychiatric condition. Chronic pain condition other than FM.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 2 months
  Pain intensity

SECONDARY OUTCOMES:
Use of rescue medication | 2 months
Visual analog scales (VAS) | 2 months
  Changes in levels of patients' pain unpleasantness, fatigue, sleep quality, mood and mental confusion.
Fibromyalgia Impact Questionnaire | 2 months
Profile of Mood States (POMS) | 2 months
Multidimensional Fatigue Inventory (MFI-20) | 2 months
Beck Depression Inventory (BDI) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Shir, MD, Principal Investigator — MUHC - Research Institute
Locations (1):
- Montreal General Hospital - Alan Edwards Pain Management Unit, Montreal, Quebec, Canada